CLINICAL TRIAL: NCT00753298
Title: A Multi-centre, Double-blind, Randomized, Parallel Groups Study Comparing PVC and Polyolefin-based Elastomer (POBE) as Catheter Materials, Outcomes Will be Measured by Subject Perception.
Brief Title: A Randomized, Fully-blinded Parallel Groups Study of Catheter Materials Used for Clean Intermittent Catheterisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YA-CLO-0002
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2012-09

CONDITIONS: Urinary Catheterization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LoFric Primo (POBE) single-use urinary catheter (Experimental)
  Interventions: Device: LoFric Primo (POBE) single-use urinary catheter
- LoFric Primo (PVC) single-use urinary catheter (Active Comparator)
  Interventions: Device: LoFric Primo (PVC) single-use urinary catheter

INTERVENTIONS:
Device: LoFric Primo (POBE) single-use urinary catheter — LoFric Primo (POBE) single-use urinary catheter
  Arms: LoFric Primo (POBE) single-use urinary catheter
Device: LoFric Primo (PVC) single-use urinary catheter — LoFric Primo (PVC) single-use urinary catheter
  Arms: LoFric Primo (PVC) single-use urinary catheter

SUMMARY:
The study is designed as a randomized, double-blind, parallel-group, multi centre study comparing perception and tolerability of investigational product and comparator. In the randomized part of the study the subjects will be given either LoFric Primo (POBE) or the comparator LoFric Primo (PVC) for use over 4 weeks. The hypothesis is that subject perception and satisfaction of POBE is equal to or better than for PVC.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Males and females aged 18 years and over
* Experienced users of LoFric Primo with a minimum of one month of use
* Practice CIC with LoFric Primo at least 3 times per day
* Adults able to read, write and understand information given to them regarding the study

Exclusion Criteria:

* Ongoing symptomatic UTI
* Suspicions of possible poor compliance with CIC during the study period
* Previous enrolment or randomisation of treatment in the present study
* Pregnancy
* Subjects not able to perform self-catheterisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred J Witjes, Prof Dr, Principal Investigator — Radboud Univesity Nijmegen Medical Centre
Locations (13):
- Medical University of Vienna, Department of Urology, Vienna, Austria
- Germany (3):
  - NRZ Greifswald, Greifswald
  - Kliniken Maria Hilf GmbH, Zentrum für Kontinenz und Neuro-Urologie, Krankenhaus St. Franziskus, Mönchengladbach
  - BG-Klinik Tübingen, Tübingen
- Italy (2):
  - Ospedale Careggi, Unità Spinale, Florence
  - Primario U.O. Neuro-Urologia, Direttore Dipartimento delle Mielolesioni, Torino
- Netherlands (4):
  - Ziekenhuis Lievensberg, Afdeling Urologie, Bergen op Zoom
  - Albert Schweitzer Ziekenhuis, Locatie Dordwijk, Dordrecht
  - Catharina Ziekenhuis, Eindhoven
  - Radboud Univesity Nijmegen Medical Centre, Nijmegen
- Verksamhet Urologi, Sahlgrenska Universitets sjukhuset, Gothenburg, Sweden
- United Kingdom (2):
  - Sheffield Teaching Hospitals NHS Foundation trust, Royal Hallamshire Hospital, Sheffield
  - Royal National Orthopaedic Hospital, Spinal Injuries Unit, Brockley Hill Stanmore, Stanmore

RESULTS

PARTICIPANT FLOW:
Groups:
- LoFric Primo (POBE): LoFric Primo (POBE) single-use urinary catheter (Arm A)
- LoFric Primo (PVC): LoFric Primo (PVC) single-use urinary catheter (Arm B)
Period: Overall Study
Arm/Group | LoFric Primo (POBE) | LoFric Primo (PVC)
Started | 97 | 98
Completed | 89 | 94
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LoFric Primo (POBE) | LoFric Primo (PVC) | Total
Number analyzed (Participants) | 97 | 98 | 195
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 74 | 148
  >=65 years | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (16.16) | 51.1 (17.20) | 52 (16.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 19 | 44
  Male | 72 | 79 | 151
Region of Enrollment [Number; unit: participants]
  Austria | 16 | 18 | 34
  Germany | 22 | 20 | 42
  Netherlands | 22 | 22 | 44
  United Kingdom | 2 | 1 | 3
  Italy | 21 | 23 | 44
  Sweden | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Subject's Perception Regarding Handling of Test Catheter Before Insertion
Description: Subject's perception regarding handling of test catheter before insertion, measured by mean score on a scale from 1 (Easy) to 5 (Troublesome)
Time Frame: At 4 weeks
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | LoFric Primo (POBE) | LoFric Primo (PVC)
Number analyzed (Participants) | 89 | 94
Score on scale | 1.71 (1.13) | 1.76 (1.05)

2. Primary Outcome: Subject's Perception Regarding Handling of Test Catheter at Insertion
Description: Subject's perception regarding handling of test catheter at insertion, measured by mean score on a scale from 1 (Easy) to 5 (Troublesome)
Time Frame: At 4 weeks
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | LoFric Primo (POBE) | LoFric Primo (PVC)
Number analyzed (Participants) | 89 | 94
Score on scale | 1.81 (1.23) | 1.55 (0.84)

3. Primary Outcome: Subject's Perception Regarding Handling of Test Catheter at Withdrawal
Description: Subject's perception regarding handling of test catheter at withdrawal, measured by mean score on a scale from 1 (Easy) to 5 (Troublesome)
Time Frame: At 4 weeks
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | LoFric Primo (POBE) | LoFric Primo (PVC)
Number analyzed (Participants) | 89 | 94
Score on scale | 1.55 (0.93) | 1.44 (0.77)

4. Primary Outcome: Subject's Perception Regarding Handling of Test Catheter After Withdrawal
Description: Subject's perception regarding handling of test catheter after withdrawal, measured by mean score on a scale from 1 (Easy) to 5 (Troublesome)
Time Frame: At 4 weeks
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | LoFric Primo (POBE) | LoFric Primo (PVC)
Number analyzed (Participants) | 89 | 94
Score on scale | 1.63 (1.05) | 1.69 (0.98)

5. Primary Outcome: Subject's General Satisfaction With Test Catheter
Description: Subject's general satisfaction with test catheter, measured by mean score on a scale from 1 (Very satisfied) to 5 (Absolutely not satified)
Time Frame: At 4 weeks
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | LoFric Primo (POBE) | LoFric Primo (PVC)
Number analyzed (Participants) | 89 | 94
Score on scale | 2.01 (0.99) | 1.75 (0.68)

6. Primary Outcome: Subject's Sensation When Using Test Catheter
Description: Subject's sensation when using test catheter, measured by mean score on a scale from 1 (Comfortable) to 6 (Severe pain)
Time Frame: At 4 weeks
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | LoFric Primo (POBE) | LoFric Primo (PVC)
Number analyzed (Participants) | 89 | 94
Score on scale | 1.86 (0.90) | 1.91 (0.92)

ADVERSE EVENTS:
Arm/Group | LoFric Primo (POBE) | LoFric Primo (PVC)
Serious Adverse Events (participants affected / at risk) | 2/97 | 1/98
Other Adverse Events (participants affected / at risk) | 3/97 | 7/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LoFric Primo (POBE) (N=97) | LoFric Primo (PVC) (N=98)
Hospitalization due to neurological problems (Nervous system disorders) | 1 | 0
Sepsis due to Urinary Tract Infection (Blood and lymphatic system disorders) | 0 | 1
Pseudotumor cerebri (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LoFric Primo (POBE) (N=97) | LoFric Primo (PVC) (N=98)
Urinary Tract Infection (Renal and urinary disorders) | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Astra Tech shall have a period of 30 days from receipt of the proposed final manuscript for any publication or other disclosure to review it and may within such time require that submission for publication or disclosure of the manuscript be delayed in order for Astra Tech to file patent applications.